CLINICAL TRIAL: NCT01442922
Title: Intervertebral Disc Nucleus Augmentation With Allograft Meniscus With Minimally Invasive Surgical Procedure
Brief Title: Intervertebral Disc Augmentation With Minimally Invasive Surgical Procedure
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 37-2011
Record Dates: First submitted 2011-09-23; First posted 2011-09-29 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2012-12

CONDITIONS: Degenerative Disc Disease
Keywords: L3-L4; L4-L5; L5-S1; Human Meniscus Allograft; Nucleus pulposus; Minimally invasive surgery; Degeneration of L3-L4 Intervertebral Disc; Degeneration of L4-L5 Intervertebral Disc; Degeneration of L5-S1 Intervertebral Disc
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human Meniscus Allograft (HMA): Patients with degenerative disk disease at L3-L4, L4-L5, or L5-S1 scheduled to undergo surgery for (HMA) implantation to replace the nucleus pulposus.
  Interventions: Other: completion of the (VAS) for level of back pain; Other: completion of the (OLBPQ) for assessment of function

INTERVENTIONS:
Other: completion of the (VAS) for level of back pain — Patients will complete the (VAS) pre-operatively and post-operatively at 6 wks, and 3, 6, 12, and 24 mos.
Other: completion of the (OLBPQ) for assessment of function — Patients will complete the (OLBPQ) pre-operatively and post-operatively at 6 wks, and 3, 6, 12, and 24 mos.

SUMMARY:
The primary purpose of the study is to establish the degree and duration of pain relief following minimally invasive surgery for a painful degenerative disc.

DETAILED DESCRIPTION:
The investigators will study patient recovery (outcome measures) in patients who have had minimally invasive surgery for implantation of human meniscus allograft (HMA) to replace the nucleus pulposus of a degenerative intervertebral disc.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of degenerative disk disease at L3-L4, L4-L5, or L5-S1
* low back for no more that one year prior to enrollment

Exclusion Criteria:

* Osteoporosis
* Degenerative changes of vertebral endplates (obvious fractures, osteophytes)
* Modic Type II changes indicative of advanced bony degeneration
* Facet arthrosis (loss of facet joint cartilage, increased synovial fluid collection, or presence of osteophytes in inferior or superior plates)
* Discs classified with stage I or II degeneration
* Patients unable to have an MRI (pacemaker, claustrophobia, etc.)

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with degenerative disk disease at L3-L4, L4-L5, or L5-S1 scheduled to undergo surgery for HMA implantation to replace the nucleus pulposus.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) documentation of the level of back pain. The (VAS) will describe the change in the level of back pain from the pre-op level. | Patients will complete the (VAS) at pre-op and at 6 wks. and at 3, 6, 12, and 24 mos. post-operatively.
  Patients will complete the (VAS) pre-operatively and post-operatively at 6 wks, and 3, 6, 12, and 24 mos. Responses are expressed on a ten centimeter line, with 0 representing no pain and 10cm representing the worst pain possible. The patient places a mark across the line representing where their perceived pain lies, from no pain to severe pain.

SECONDARY OUTCOMES:
The Oswestry Low Back Pain Disability Questionnaire (OLBPQ) function assessment The (OLBPQ) will describe the change in the level of function from the pre-op level. | Patients will complete the (OLBPQ) at pre-op and at 6 wks. and at 3, 6, 12, and 24 mos. post-operatively.
  Patients will complete the (OLBPQ) pre-operatively and post-operatively at 6 wks, and 3, 6, 12, and 24 mos. This is a 10-question self-rating scale used to evaluate the degree of functional impairment a patient is experiencing in a number of activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mac Millan, M.D., Principal Investigator — University of Florida Department of Orthopaedics and Rehabilitation
Locations (1):
- UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States